CLINICAL TRIAL: NCT05806554
Title: Accuracy and Precision of the True Vie I3 Continuous Glucose Monitoring System: an Open Label, Multi-Center Trial
Status: Completed | Type: Observational
Sponsor: Sinocare (Industry)
Collaborators: Integrated Medical Development (Industry)
Responsible Party: Sponsor
Other Study IDs: NPI031-CIP-002F
Record Dates: First submitted 2023-03-28; First posted 2023-04-10 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (2):
- T1DM: Participants with type 1 diabetes mellitus
  Interventions: Device: Continuous glucose monitoring device
- T2DM: Participants with type 2 diabetes mellitus
  Interventions: Device: Continuous glucose monitoring device

INTERVENTIONS:
Device: Continuous glucose monitoring device — Continuous glucose monitoring device

SUMMARY:
The purpose of the investigation is to evaluate the performance of the I3 CGM according to the FDA's special controls for iCGM.

DETAILED DESCRIPTION:
Participants will attend a screening visit, 4 clinic visits with Frequent Sampling Testing (FST) at the beginning, 2 in the middle, and end of the I3 CGM sensor wear, and a visit for removal of the I3 CGM. Participants will wear 3 I3 CGM devices for up to 15 days and be instructed to continue their normal daily activities and manage their glucose as usual between in clinic FST per routine care. Participants will not have access to the I3 CGM data for the management of their blood glucose between clinic visits and will continue their usual care including CGM, if they are CGM users.

At the clinic FST visits venous blood samples will be drawn from an intravenous cannula for FST for up to 10 hours for plasma glucose determination. During the clinic visits the investigative site staff will determine the participants' insulin doses and meals and may induce both hypoglycemia and hyperglycemia of up to an hour duration.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with T1DM or T2DM diagnosed for at least 6 months. 2. Individual is 18-80 years old, inclusive, at the time of screening. 3. Must be and have been in stable treatment regimen for at least 1 month with a multiple daily insulin dosing regimen (at least two insulin doses with meals daily) or CSII using at least two bolus doses a day with meals, irrespective of delivery device(s).

Exclusion Criteria:

* 1. History of skin adhesive tolerance issues in the area of sensor placement. 2. HbA1c > 9%. 3. Insulin meal dosing based on fixed dose regimens. 4. Absence of established correction factor for high glucose. 5. Hematocrit below 10% under the lower limit of the normal range. 6. Body mass index < 18.5 kg/m2. 7. Inadequate intravenous access on arms. 8. Participant has had a hypoglycemic seizure within the past 6 months prior to enrollment.

  9. Participant has had an episode of diabetic ketoacidosis (DKA) within the past 6 months prior to enrollment.

  10. Participant has a history of a seizure disorder. 11. Pregnancy, planned pregnancy within the study period, or unwillingness to use reliable contraception during the study period.

  12. Planned MRI, CT scan or diathermia procedure for the duration of the study.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with type 1 diabetes mellitus (T1DM) or type 2 diabetes mellitus (T2DM) using an insulin treatment regimen based on carbohydrate (CHO) counting for meal insulin dose determination and 18-80 years of age will be recruited to participate in the study. Both participants using and not using CGM will be recruited, and participants with a wide range of BMIs and ages will be represented.
Sampling Method: Non-Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2023-07-19 (Actual); Primary Completion 2024-06-13 (Actual); Study Completion 2024-10-22 (Actual)

PRIMARY OUTCOMES:
Accuracy | 15 days
  percentage of iCGM values in the measuring range less than 70 mg/dL (3.9 mmol/l) within +/- 15 mg/dL (0.83 mmol/l) of the

CONTACTS AND LOCATIONS:
Overall Officials: Ron Brazg, MD, Principal Investigator — RCRC
Locations (6):
- United States (4):
  - Woodland Research Northwest, Rogers, Arkansas
  - Diablo Clinical Research, Walnut Creek, California
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Rainier Clinical Research Center, Renton, Washington
- Germany (2):
  - PSHI Praxis GmbH, Mainz
  - Institut für Diabetes-Technologie Forschungs- und Entwicklungsgesellschaft mbH an der Universität Ulm, Ulm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jendrike N, Link M, Oter S, Fei J, Zheng J, Gao F, Gao A, Zhu S, Shi L, Strange P, Flacke F, Eichenlaub M, Freckmann G. Performance of a New Continuous Glucose Monitoring System in German Adults Living with Diabetes. Diabetes Ther. 2025 Dec 29. doi: 10.1007/s13300-025-01832-6. Online ahead of print. PMID 41461989